CLINICAL TRIAL: NCT02838290
Title: Occupational Distress in Doctors: The Effect of an Induction Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birkbeck, University of London (Other)
Responsible Party: Principal Investigator, Asta Medisauskaite, Doctoral Researcher, Birkbeck, University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01N/A
Record Dates: First submitted 2016-06-06; First posted 2016-07-20 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Burnout, Professional; Anxiety; Grief; Adaptation, Psychological; Eating Behavior; Alcohol Drinking; Drug Use
Keywords: Burnout; Psychiatric morbidity; Anxiety; Grief; Alcohol and drug use
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Feeding Behavior; Alcohol Drinking; Burnout, Psychological | interventions — Neoadjuvant Therapy; Control Groups

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Induction (Experimental)
  Interventions: Other: Induction
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Induction — Participants will be randomly assigned (computer generated straight away after clicking the link to the research) to one of 4 experimental conditions: stress at work, dealing with a patient's death, managing stress at work or all topics together. Each module includes brief reflection parts and quizzes. Participants will be asked to fill in an online survey just before the induction and a week after. The survey is about current occupational distress and organizational factors.
  Arms: Induction
Other: Control group — Participants in the control group will be asked to fill in an online survey, but will not have any task at time-1. However, participants in the control group will be invited to complete induction programme after time-2 (a week time after time-1) in ensure the same expectations in both, experimental and control, groups.
  Arms: Control group

SUMMARY:
Background: Over 39% of approximately 3,000 doctors (The British Medical Association quarterly survey, 2015) admitted to frequently feeling drained, exhausted, overloaded, tired, low and lacking energy. Such occupational distress may link to psychological and physical difficulties in doctors and have negative outcomes for organization and patients. The aim of the current study is to investigate the impact of an induction programme on occupational distress of doctors.

Methods/design: Doctors will be invited to take part in an online research. Participants will be randomly assigned to the experimental and control groups. Participants in the experimental groups will complete one of the induction topics (about stress at work). Before and after an induction programme participants will be asked to fill in an online survey about their current occupational distress and organizational well-being.

Discussion: The investigators expect that doctors' psychological, physiological and organizational well-being will improve after an induction programme which should serve as a resource for better doctor's own health understanding.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors across all specialties and professional grades who have a regular contact with patients and works in the United Kingdom.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The Anxiety Disorder Scale | A week
The Grief Inventory | A week
The Coping Mechanisms Scale | A week
  Self-distraction, active coping, substance use, use of emotional support, use of instrumental support, positive reframing, humour, self-blame
The Psychiatric Morbidity Scale | A week
The Physical Symptoms Scale | A week
The Insomnia Scale | A week
The Binge Eating Scale | A week
The Burnout Inventory | A week
Alcohol use | A week
Drug use | A week

SECONDARY OUTCOMES:
The Effort-Reward Scale | A week
The Work Engagement Scale | A week
The Work-Family Conflict Scale | A week

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medisauskaite A, Kamau C. Does occupational distress raise the risk of alcohol use, binge-eating, ill health and sleep problems among medical doctors? A UK cross-sectional study. BMJ Open. 2019 May 15;9(5):e027362. doi: 10.1136/bmjopen-2018-027362. PMID 31092661
- [Derived] Medisauskaite A, Kamau C. Reducing burnout and anxiety among doctors: Randomized controlled trial. Psychiatry Res. 2019 Apr;274:383-390. doi: 10.1016/j.psychres.2019.02.075. Epub 2019 Mar 1. PMID 30852432